CLINICAL TRIAL: NCT01358006
Title: An Open Label Dose-Ranging Study in Healthy Male Subjects to Investigate the Binding Potential of JNJ-40411813 to Serotonin 2A Receptors in the Central Nervous System
Brief Title: A Dose-Ranging Study of JNJ-40411813 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR017485; 40411813EDI1008 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2010-022176-32 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: JNJ-40411813; Positron Emission Tomography (PET); Serotonin-2A (5-HT2A) receptor antagonist; Male Volunteers
MeSH Terms: interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): JNJ-40411813 Cohort 1: Type=2 to 3 unit=mg number=200 to 300 form=capsule route=oral use.Capsule(s) taken in the fed state Capsule(s) taken in the fed state.,JNJ-40411813 Cohort 2: Type=up to 7 unit=mg number=up to 700 mg form=capsule route=oral use. Capsule(s) taken in the fed state.
  Interventions: Drug: JNJ-40411813

INTERVENTIONS:
Drug: JNJ-40411813 — Cohort 1: Type=2 to 3, unit=mg, number=200 to 300, form=capsule, route=oral use.Capsule(s) taken in the fed state Capsule(s) taken in the fed state.
Drug: JNJ-40411813 — Cohort 2: Type=up to 7, unit=mg, number=up to 700 mg, form=capsule, route=oral use. Capsule(s) taken in the fed state.

SUMMARY:
The purpose of this study is to characterize the 5-HT2A binding over the maximum feasible dose range of JNJ-40411813, to estimate the plasma concentration associated with 50% 5-HT2A binding, and to investigate the safety and tolerability of JNJ-40411813 in healthy male volunteers.

DETAILED DESCRIPTION:
This will be an open-label (volunteers and study staff will know the identity of assigned treatment), dose-ranging study to determine 5-HT2A receptor engagement by JNJ-40411813 as a function of dose and time in healthy male volunteers. The study will consist of an eligibility screening examination, an open-label treatment period and a follow-up examination (approximately 10 days after dose administration, a follow-up examination will be performed). Initially, 4 volunteers (Cohort 1) will be included to determine 5-HT2A receptor occupancy following single dose administration of JNJ-40411813. Dependent on the results, doses for the remaining 8 volunteers (Cohort 2 and 3) will be selected to further characterize 5-HT2A receptor occupancy within the feasible dose range up to maximally 700 mg JNJ-40411813.The maximal study duration for a volunteer will be 6 weeks. In this study, [11C]-MDL 100,907 will be used as positron emission tomography (PET) ligand to investigate the concentration-related binding of 40411813 to the 5-HT2A receptor in the brain. JNJ-40411813 (200 mg to 700 mg) will be taken orally (by mouth). If multiple capsules have to be taken, the actual intake may be spread over a 15-minute period. Study drug will be administered to each volunteer just after completion of a meal and within 30 minutes after the start of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kg/m2, inclusive
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Volunteers must sign an informed consent to document that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Have abnormal values for clinical laboratory tests, clinically significant abnormal physical examination findings, vital signs, or 12-lead Electrocardiograms (ECGs) performed at screening considered to be of clinical significance to the Investigator
* Have Significant history of or current significant medical illness that the Investigator considers should exclude the volunteer
* Have known allergies, hypersensitivity, or intolerance to JNJ-40411813, its excipients, or to the PET ligand used in the study
* Have significant history of psychiatric or neurological illness in first-degree relatives
* Been exposed to ionizing radiation as a volunteer (including diagnostic procedures)
* Presence of other exclusion criteria as specified in the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
5-HT2A binding determined by Positron Emission Tomography (PET) scans | Up to 24 hours after study drug administration

SECONDARY OUTCOMES:
Plasma concentration of JNJ-40411813 | Up to 2 days
Adverse Events Reported | Up to 10 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Groningen, Netherlands